CLINICAL TRIAL: NCT04382677
Title: Intervention to Improve Outcomes for Foster Children Reunited With Their Birth Families
Brief Title: Families Together: Intervention for Reunified Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Monica Oxford, Research Professor: School of Nursing, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-110816-S; R01HD090176 (NIH)
Record Dates: First submitted 2020-04-28; First posted 2020-05-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Child Abuse; Child Neglect
Keywords: Child Welfare; Child Protective Services; Parenting
MeSH Terms: interventions — Health Resources; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Promoting First Relationships (Experimental): The PFR program designed for birth families being reunited after foster care placement consists of a manualized 12-session intervention delivered in the home by trained providers.
  Interventions: Behavioral: Promoting First Relationships ®
- Resource & Referral (Other): The service consists of a needs assessment conducted by phone, followed by a personalized resource packet and referrals, and 3 monthly check-in phone calls.
  Interventions: Other: Resource & Referral

INTERVENTIONS:
Behavioral: Promoting First Relationships ® — Promoting First Relationships ® is based on attachment theory and is strengths-based. The 12 week intervention is delivered in the home of the family. Each week has a theme for discussion, handouts, an activity, and time for "joining" - checking in with the parent, listening to their concerns, and establishing a positive, supportive relationship. The provider videotapes playtime between parent and child, and alternates weeks watching the video with the parent, reflecting about the needs of both parent and child (reflective observation). PFR consultation strategies include Joining, Positive Feedback, Instructive Feedback, Reflective Questions and Comments, and Instruction with Handouts. These core strategies enhance parents' sense of security and competency. The provider helps the parent develop greater empathy and understanding of the child's needs and feelings, and helps the parent to identify their own feelings and needs around parenting.
  Other Names: PFR
  Arms: Promoting First Relationships
Other: Resource & Referral — This condition consists of 1) Resource & Referral assistance provided over the phone, and 2) Local Services Resource Packet. Throughout the intervention period, the provider makes monthly phone calls to offer further support to families, answer questions, and provide additional resources. The provider has at least four interactions with each family served. In addition, families in this condition have the Resource and Referral Specialist's phone number and they can call if an additional need arises. The resource packet includes local information organized by type of need or resource. These packets are updated regularly as services change over time.
  Other Names: R&R
  Arms: Resource & Referral

SUMMARY:
Birth parents of young children who have been placed into foster care are a highly vulnerable population of caregivers. Little is known about the ability of existing prevention programs to intervene with birth parents who have recently been reunified with their children under the age of six. This project aims to evaluate a brief, home-visiting intervention model with a sample of reunified birth parents, examining its effectiveness to improve parenting and child wellbeing, and reduce reoccurrence of maltreatment and reunification failure.

DETAILED DESCRIPTION:
There is no brief, home visiting, evidence-based intervention designed for and evaluated with Child Welfare System (CWS) birth parents and their children under six, once they are reunified. Why is this important? Because reunified birth parents represent one of the highest risk subpopulations of parents whose challenges contribute both to their child's exposure to stress and trauma and to the intergenerational transmission of impaired parenting, maltreatment, and foster care placement.

Reunified birth parents are more likely than other parents to have been foster children and survivors of childhood maltreatment. They have higher rates of co-morbid mental health disorders, substance abuse, poverty, low education, and homelessness. When their children are placed in out-of-home care as infants or toddlers, they are more likely to have longer stays in foster care than any other age group. Foster children are at risk for serious emotional, behavioral, neurological, and physiological health problems, and for continued relationship disruptions, maltreatment, and foster care placements throughout their life course. Birth parents need intervention services when they reunite with their child to support the already fragile parent-child relationship. Even when birth parents work hard to fulfill court requirements to regain custody of their child, they are often left without the skills necessary to establish a strong and lasting connection with their child. This failure of service, we believe, leads reunified families to experience a high rate of maltreatment reoccurrence and reentry into foster care.

In this application we will evaluate the effectiveness of a community based, home visiting intervention program with a population of birth parents recently reunified with their child under the age of six after a foster care placement. In order to do this, we first adapt the program by adding material relevant to reunified birth families and adapt the material for older children. We will evaluate the effectiveness of Promoting First Relationships ® (PFR; Kelly et al., 2008) to meet the parenting needs of this vulnerable population. Promoting First Relationships was originally designed for children birth to three, and we will expand the curriculum to meet the needs of children through age six. Through a strong, established community partnership between the state, a community mental health agency, and the University of Washington, we will 1) adapt Promoting First Relationships ® (PFR) for reunified birth families and older children; 2) test the effectiveness of PFR to improve parental quality and parent-child interaction as compared to a Resource and Referral service; 3) test the effectiveness of PFR on reducing social, emotional, and behavioral problems in a population of children at risk for elevated emotional and behavioral disorders; 4) test the effectiveness of PFR in reducing referrals to Child Protective Services (CPS) and re-entry into foster care; and 5) test a proposed PFR theoretical model, linking the PFR intervention to improved parental insightfulness and emotional competence, which then contributes to parental sensitivity and improved child outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Birth parents reunited with their child (age 1-5 years) after a foster or kin care placement in trial return home status
* Parenting the child at study enrollment
* Child Welfare case served by the following Washington State offices: all of Region 2 South, Lynnwood, Tacoma, Everett, Smokey Point, and Lakewood
* Birth parents must be age 18 or older, mothers and fathers are eligible (one parent per study child enrolled)
* Conversant in English
* Access to a telephone
* Housing situation allows for home visits

Exclusion Criteria:

* Experiencing an acute crisis (e.g., hospitalization, incarceration)
* Previously received the Promoting First Relationships ® intervention or Child Parent Psychotherapy (CPP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Child Welfare Services removal from birth parent home | 1 year post intervention
  Official child welfare administrative records indicating whether child was removed from the birth parent home.
Change in Parental Sensitivity (Video recorded observations coded by coders blind to intervention) | Post intervention (Time 2) -- approximately 6 months after Baseline (Time 1)
  Parent sensitivity is measured by the Nursing Child Assessment Teaching Scale (NCATS;Barnard 1994), a videotaped interaction to assess caregiver sensitivity, stimulation of the child, and emotional responsiveness during interaction. The score is the sum of 50 items, ranging from 0 to 50; higher scores indicate greater parental sensitivity.
Change in Parental Sensitivity (Video recorded observations coded by coders blind to intervention) | 6 months post intervention (Time 3) -- approximately 12 months after Baseline (Time 1)
  Parent sensitivity is measured by the Nursing Child Assessment Teaching Scale (NCATS;Barnard 1994), a videotaped interaction to assess caregiver sensitivity, stimulation of the child, and emotional responsiveness during interaction. The score is the sum of 50 items, ranging from 0 to 50; higher scores indicate greater parental sensitivity.
Change in Parenting Knowledge of Child Development | Post intervention (Time 2) -- approximately 6 months after Baseline (Time 1)
  21-item Likert-scale questionnaire developed by study, "Raising a Child". The score is the mean ranging from 1 to 4; higher scores indicate greater parenting knowledge.
Change in Parenting Knowledge of Child Development | 6 months post intervention (Time 3) -- approximately 12 months after Baseline (Time 1)
  21-item Likert-scale questionnaire developed by study, "Raising a Child". The score is the mean ranging from 1 to 4; higher scores indicate greater parenting knowledge.

SECONDARY OUTCOMES:
Change in Child Externalizing Problem Behavior | Post intervention (Time 2) -- approximately 6 months after Baseline (Time 1)
  Child externalizing behavioral problems will be measured based on parent report using the Child Behavior Check List (CBCL: Achenbach & Rescorla, 2000). The externalizing scale has 24 items; raw scores can range from 0 to 48 with higher scores indicating more externalizing behaviors.
Change in Child Externalizing Problem Behavior | 6 months post intervention (Time 3) -- approximately 12 months after Baseline (Time 1)
  Child externalizing behavioral problems will be measured based on parent report using the Child Behavior Check List (CBCL: Achenbach & Rescorla, 2000). The externalizing scale has 24 items; raw scores can range from 0 to 48 with higher scores indicating more externalizing behaviors.
Change in Child Internalizing Problem Behavior | Post intervention (Time 2) -- approximately 6 months after Baseline (Time 1)
  Child internalizing behavioral problems will be measured based on parent report using the Child Behavior Check List (CBCL: Achenbach & Rescorla, 2000). The internalizing scale has 36 items; raw scores can range from 0 to 72 with higher scores indicating more internalizing behaviors.
Change in Child Internalizing Problem Behavior | 6 months post intervention (Time 3) -- approximately 12 months after Baseline (Time 1)
  Child internalizing behavioral problems will be measured based on parent report using the Child Behavior Check List (CBCL: Achenbach & Rescorla, 2000). The internalizing scale has 36 items; raw scores can range from 0 to 72 with higher scores indicating more internalizing behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Monica L Oxford, MSW, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Child, Family, and Population Health Nursing, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No